CLINICAL TRIAL: NCT05569382
Title: Treatment Effects of Bisoprolol and Verapamil in Symptomatic Patients With Non-obstructive Hypertrophic Cardiomyopathy
Acronym: TEMPO II
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Morten Steen Kvistholm Jensen (Other)
Collaborators: Viborg Regional Hospital (Other); Zealand University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Morten Steen Kvistholm Jensen, Consultant, PhD, Associated professor, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 490-73-6795; 2021-006953-77 (EudraCT Number)
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Non-obstructive Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy; Bisoprolol; Verapamil; Beta Blocker; Calcium-channel Blocker
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Verapamil; Bisoprolol

STUDY DESIGN:
Intervention Model Description: The trial will be performed and analyzed in three phases, and each phase may be unblinded and analyzed separately.
  Phase one: More than 26 patients must have completed all three treatment periods. Functional analyses of VO2 max from CPX tests and secondary functional effect parameters (KCCQ, NYHA, CCS), echocardiographic parameters, biomarkers (TNI/TNT, pro-BNP/BNP).
  Phase two: Between 30 to 50 patients must have completed all three treatment periods and have CMR performed in each period. Structural and hemodynamic analyses of cardiac dimensions and hemodynamic effect parameters (CMR). Sex specific analyses of functional, structural and hemodynamic effect parameters will be performed.
  Phase three (n > 82): Arrhythmic effect parameters will be analyzed from ambulatory ECG monitoring.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verapamil (Active Comparator): Maximal tolerable dose (up to 360 mg per day)
  Interventions: Drug: Verapamil
- Bisoprolol (Active Comparator): Maximal tolerable dose (up to 7,5 mg per day)
  Interventions: Drug: Bisoprolol
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verapamil — 1. week: uptitration with 120 mg capsules per day, until maximum dosage of 360 mg´s/day.
  2-4. week: steady state treatment with the maximum tolerated dose.
  5. week: downtitration
  Other Names: Isoptin Retard 240 MG; Verapamil Hydrochloride 240 MG
  Arms: Verapamil
Drug: Bisoprolol — 1. week: uptitration with 2.5 mg capsules per day, until maximum dosage of 7.5 mg´s/day.
  2-4. week: steady state treatment with the maximum tolerated dose.
  5. week: downtitration
  Other Names: Bisoprolol "Krka" 2.5 MG; Bisoprolol Fumarate 2.5 MG
  Arms: Bisoprolol
Drug: Placebo — 1. week: uptitration with one capsules per day, until maximum dosage of three capsules/day.
  2-4. week: steady state treatment with the maximum tolerated dose.
  5. week: downtitration
  Other Names: Placebo oral capsule
  Arms: Placebo

SUMMARY:
Aim: to compare the treatment effects of Bisoprolol (beta 1 receptor specific beta blocker (BB)) and Verapamil (cardio-specific calcium channel blockers (CCB)) in patients with non-obstructive hypertrophic cardiomyopathy (HCM).

Background: Hypertrophic cardiomyopathy (HCM) is characterized by hypertrophy of the left ventricular wall and a hypercontracted state of the sarcomeres. This narrows the left ventricular cavity, but though the left ejection fraction is increased the stroke volume and the cardiac output cannot be fully compensated. The disease manifestations can be mild or develop into severe functional limitations and devastating complications at early age. Dyspnea, chest pain, palpitations and syncope are the most common symptoms, and patients are at risk of supraventricular and ventricular arrhythmias. Arrhythmias and sudden cardiac deaths may precede heart failure symptoms. Patients with symptomatic HCM are treated initially with beta blockers and calcium channel blockers. However, there is limited evidence supporting the effectiveness of this guideline-recommended treatment in HCM.

Methods: The study is a multicenter, double-blinded, randomized, placebo-controlled cross-over trial. Patients are randomized in to three 35-days treatment periods with Bisoprolol, Verapamil and Placebo. Each treatment period includes a 7-days up titration period, a 21-days target dose period and a 7-days down titration period. Between treatment periods 45 days treatment pause is allowed. End point will be evaluated at day 21 (- 4 days). Patients will be evaluated by cardiopulmonary exercise test, echocardiography, 7 day Holter-monitoring, biomarkers and the Kansas City Cardiomyopathy Questionnaire (KCCQ). A subgroup of patients will also be evaluated with cardiac magnetic resonance imaging.

Hypotheses: Three separate phases each with one primary effect parameters will be analyzed between treatment with Bisoprolol and Verapamil:

Phase 1: The maximal oxygen consumption (VO2 max) is different (ΔVO2 max ≥1 ml/kg/min) between treatments in non-obstructive HCM patients Phase 2: The left ventricular enddiastolic volume (LVvol) is different (ΔLVvol ≥3 ml) between treatments in non-obstructive HCM patients.

Phase 3: The incidence of non-sustained ventricular tachycardia (NSVT) is different (Hazard ratio ≥ 0.5) between treatments in non-obstructive HCM patients.

The trial will be performed and analyzed in three phases, and each phase may be unblinded and analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Maximal wall thickness ≥ 15 mm unrelated to hypertension, valve diseases or storage diseases. And one of the following:

  1. New York Heart Association - functional class (NYHA) ≥ II
  2. A history of NYHA class ≥ II before treatment with BB or CCB
  3. Pro-BNP>300 ng/l/35>nmol/l or BNP >100ng/l/>29nmol/l
  4. Non-sustained VT (>120 min-1, ≥3 cycles) documented within the last 2 years of screening

Exclusion Criteria:

* Left ventricular ejection fraction < 50%
* LVOT gradient >30 mmHg at rest or during Valsalva maneuver after discontinuation of BB or CCB respectively
* History of LVOT gradient >30 mmHg at rest, during exercise or during Valsalva maneuver.
* Permanent atrial fibrillation
* Permanent right ventricular pacing
* Previous intolerance for Bisoprolol (BB) or Verapamil (CCB)
* Known present obstructive coronary disease (previous percutaneous coronary intervention is accepted)
* eGFR < 40 ml/min
* Fertile women (<50 years) who are pregnant (Positive Plasma-HCG), breastfeeding or not using anticonception.
* Significant liver failure
* Severe valvular disease
* Bradycardia (40bpm)
* Hypotension (systolic <100mmHg)
* Other significant comorbidity or risks associated with discontinuation of BB or CCB after individual judgement by the investigators.
* Unable to understand patient information intellectually or linguistically
* Unable to perform exercise test.
* Unable to speak and/or understand Danish.

Additional exclusion criteria for CMR sub study:

* Implantable cardioverter defibrillator (any kind)
* Pacemaker (any kind)
* Metal implants like to affect image quality
* Metal implants that poses a risk during CMR
* Inability to cope with being in the scanner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO2 max) | Changes will be evaluated at day 21 in each treatment arm
  Changes in VO2 max estimated during cardiopulmonary exercise test
Left ventricular enddiastolic volume (LVvol) | Changes will be evaluated at day 21 in each treatment arm
  Changes in enddiastolic volume (LVvol) estimated during cardiac MRI
Incidence of non-sustained ventricular tachycardia (NSVT | Changes will be evaluated at day 21 +7 days in each treatment arm
  Changes in NSVT estimated during ECG monitoring

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Changes will be evaluated at day 21 in each treatment arm
  Changes in KCCQ assessed by clinical evaluation
New York Heart Association (NYHA) functional classification | Changes will be evaluated at day 21 in each treatment arm
  Changes in NYHA class assessed by clinical evaluation
Canadian Cardiovascular Society (CCS) class | Changes will be evaluated at day 21 in each treatment arm
  Changes in CCS class assessed by clinical evaluation
Pro-BNP/BNP | Changes will be evaluated at day 21 in each treatment arm
  Changes in level of Pro-BNP/BNP in blood sample
High sensitive Troponin I/Troponin T | Changes will be evaluated at day 21 in each treatment arm
  Changes in level of high sensitive Troponin I/Troponin T in blood sample
Metabolic equivalent of task (METs) | Changes will be evaluated at day 21 in each treatment arm
  Changes in METs measured during cardiopulmonary exercise test
Recovery time | Changes will be evaluated at day 21 in each treatment arm
  Changes in recovery time measured during cardiopulmonary exercise test
VO2 max Anaerobic threshold | Changes will be evaluated at day 21 in each treatment arm
  Changes in VO2 max at anaerobic threshold measured during cardiopulmonary exercise test
Percent predicted VO2 max | Changes will be evaluated at day 21 in each treatment arm
  Changes in percent predicted VO2 max measured during cardiopulmonary exercise test
Ventilatory equivalent for carbon dioxide VE/VCO2 | Changes will be evaluated at day 21 in each treatment arm
  Changes in VE/VCO2 measured during cardiopulmonary exercise test
Echocardiographic left ventricular end-diastolic dimension | Changes will be evaluated at day 21 in each treatment arm
  Changes in left ventricular end-diastolic dimension measured during echocardiography
Echocardiographic global longitudinal strain (GLS) for LV function | Changes will be evaluated at day 21 in each treatment arm
  Changes in GLS measured during echocardiography
Echocardiographic left ventricular outflow tract time velocity intergral (LVOT VTI) for LV function | Changes will be evaluated at day 21 in each treatment arm
  Changes in LVOT VTI measured during echocardiography
Echocardiographic dimension of left atrial | Changes will be evaluated at day 21 in each treatment arm
  Changes in left atrial dimension measured during echocardiography
Episodes of atrial fibrillation (AFIB) on Holter monitoring | Changes will be evaluated at day 21 +7 days in each treatment arm
  Changes in episodes of AFIB measured during Holter monitoring
Number of ventricular ectopic beats on Holter monitoring | Changes will be evaluated at day 21 +7 days in each treatment arm
  Changes in number of ventricular ectopic beats measured during Holter monitoring
Left ventricular systolic function on Cardiac MRI | Changes will be evaluated at day 21 in each treatment arm
  Changes in left ventricular systolic function on Cardiac MRI
Right ventricular dimensions on Cardiac MRI | Changes will be evaluated at day 21 in each treatment arm
  Changes in right ventricular dimensions on Cardiac MRI
Right ventricular systolic function on Cardiac MRI | Changes will be evaluated at day 21 in each treatment arm
  Changes in right ventricular systolic function on Cardiac MRI
Stroke volume (Aortic flow) on Cardiac MRI | Changes will be evaluated at day 21 in each treatment arm
  Changes in stroke volume (Aortic flow) on Cardiac MRI
Coronary sinus flow on Cardiac MRI | Changes will be evaluated at day 21 in each treatment arm
  Changes in coronary sinus flow on Cardiac MRI
Dimension of inferior and superior caval vein on Cardiac MRI | Changes will be evaluated at day 21 in each treatment arm
  Changes in dimension of inferior and superior caval vein on Cardiac MRI
Dimension of left atrium on cardiac MRI | Changes will be evaluated at day 21 in each treatment arm
  Changes in dimension of left atrium on cardiac MRI
Sex specific analyses of outcome measures | Changes will be evaluated at day 21 in each treatment arm
  Changes in outcome measures between male and female

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Department of Cardiology, Aarhus University Hospital, Aarhus N
  - Department of Cardiology, Odense University Hospital, Odense
  - Department of Cardiology, Zealand University Hospital, Roskilde
  - Department of Cardiology, Regional Hospital Viborg, Viborg